CLINICAL TRIAL: NCT06685783
Title: Vis-Rx Prime Micro-Imaging Catheter Clinical Evaluation Study
Brief Title: Vis-Rx Prime Micro-Imaging Catheter Study
Status: Active, not recruiting | Type: Observational
Sponsor: Gentuity, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: MISC-074
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To study the performance of the Gentuity® HF-OCT Imaging System and Vis-Rx Prime® Micro-Imaging Catheter when used to obtain images of coronary arteries in patients who are undergoing cardiac catheterization and are candidates for interventional procedures. The study will evaluate ease of catheter use by physicians using the catheters, image quality and overall performance. The patient's involvement in the study ends when the cardiac catheterization/interventional procedure is completed.

DETAILED DESCRIPTION:
This is a single arm, unblinded, multi-center, clinical evaluation that will be performed at 3 to 5 investigational sites in the United States with subjects who undergo HF-OCT imaging as part of their cardiac catheterization procedure. This study will evaluate a range of device operators (interventional cardiologists) as well as patients and vessels consistent with the product labeling. The operator evaluation will be determined post use of the device using a Likert Grading Scale. Clear Image Length of the acquired HF-OCT image will be measured by an independent core lab. Safety will be monitored through the interventional procedure and Adverse Events that are potentially related to either the device or the procedure will be recorded, evaluated and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Patients willing and able to provide written informed consent to participate in evaluation
* Patients who are candidates for transluminal interventional procedures for their coronary arteries (also known as PCI)

Exclusion Criteria:

* Bacteremia or sepsis
* Major coagulation system abnormalities
* Severe hemodynamic instability or shock
* Acute renal failure
* Disqualified for Coronary Artery Bypass Graft surgery
* Disqualified for Percutaneous Coronary Intervention
* Patients currently enrolled in another study to evaluate an investigational device or medication
* Any target vessel which has undergone a bypass procedure

The lesion-specific exclusion criteria assessed from angiography are:

* Total occlusion
* Coronary artery spasm
* Large thrombus (as visible under angiography)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in the cardiac catheterization lab who are candidates for PCI
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Clinical performance | During percutaneous interventional procedure
  Clinical performance of the Gentuity HF-OCT Imaging System with the Vis-Rx Prime Micro-Imaging Catheter in a real-world setting as determined by the clinical operator using a Likert Grading Scale (1-5 scale; 1=unacceptable, 5= excellent)
Technical Performance | During percutaneous interventional procedure
  Clear Image Length of the acquired HF-OCT image

OTHER OUTCOMES:
Incidence of Adverse Events | During percutaneous interventional procedure
  Adverse Events that are potentially related to either the device or the procedure

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - St. Francis Hospital and Heart Center, Roslyn, New York
  - Lindner Research Center at The Christ Hospital, Cincinnati, Ohio